CLINICAL TRIAL: NCT03283488
Title: Randomized, Double-blind Clinical Trial of the Use of Mirtazapine Versus Megestrol for the Control of Anorexia-cachexia in Cancer Patients in Palliative Care.
Brief Title: Comparison Between Mirtazapine and Megestrol for the Control of Anorexia-cachexia in Cancer Patients in Palliative Care.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Nereida Kilza da Costa Lima, Assistant Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Mirtazapine_Cachexia
Record Dates: First submitted 2017-09-10; First posted 2017-09-14 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Cachexia; Cancer; Anorexia
Keywords: anorexia; cachexia; mirtazapine; megestrol; palliative care
MeSH Terms: conditions — Cachexia; Neoplasms; Anorexia | interventions — Mirtazapine; Megestrol; Megestrol Acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mirtazapine (Experimental): Tablets of 15mg mirtazapine will be used according to randomization. At the first visit, patients will be instructed to take one tablet at night for better tolerability. From the second week, if there is good tolerance, they will take two tablets at night until the end of the study.
  Interventions: Drug: Mirtazapine
- Megestrol (Active Comparator): Tablets of 160mg megestrol will be used according to randomization. At the first visit, patients will be instructed to take one tablet at night for better tolerability. From the second week, if there is good tolerance, they will take two tablets at night until the end of the study.
  Interventions: Drug: Megestrol

INTERVENTIONS:
Drug: Mirtazapine — Tablets of 15mg mirtazapine will be used according to randomization. At the first visit, patients will be instructed to take one tablet at night for better tolerability. From the second week, if there is good tolerance, they will take two tablets at night until the end of the study.
  Other Names: Remeron
  Arms: Mirtazapine
Drug: Megestrol — Tablets of 160mg megestrol will be used according to randomization. At the first visit, patients will be instructed to take one tablet at night for better tolerability. From the second week, if there is good tolerance, they will take two tablets at night until the end of the study.
  Other Names: megestrol acetate
  Arms: Megestrol

SUMMARY:
Cancer-associated anorexia-cachexia is an insidious syndrome that has a major impact on the patient's quality of life, but is also associated with a significant reduction in survival. Despite its clinical importance, it remains a widely underestimated and untreated condition. Considering the scarcity of pharmacological measures, it is necessary to invest in studies that may contribute to the rational and effective treatment of this clinical condition. Mirtazapine has a special therapeutic potential because it is a well-tolerated drug with few adverse effects and with well-known orexigenic action in clinical practice.The objective of this study is to evaluate the effect of mirtazapine as a pharmacological measure in the management of cancer-related anorexia-cachexia in patients in palliative care. A randomized, double-blind clinical trial involving 52 cancer patients with anorexia-cachexia in palliative care will be conducted. Patients will be randomized to receive mirtazapine or megestrol and will be evaluated longitudinally for a period of 8 weeks. The primary endpoint will be to assess the effect of mirtazapine on anorexia and weight gain and secondary outcomes will be to assess the tolerability and safety of mirtazapine and the effect of mirtazapine on body composition, quality of life, and functional capacity of patients.

DETAILED DESCRIPTION:
Cancer-associated anorexia-cachexia is an insidious syndrome that has a major impact on the patient's quality of life, but is also associated with a significant reduction in survival. Unintentional weight loss can predict a poor prognosis in cancer patients which is most likely due to decreased doses of treatment. Despite its clinical importance, it remains a widely underestimated and untreated condition. Considering the scarcity of pharmacological measures, it is necessary to invest in studies that may contribute to the rational and effective treatment of this clinical condition. Mirtazapine has a special therapeutic potential because it is a well-tolerated drug with few adverse effects and with well-known orexigenic action in clinical practice. It has been shown to have side effects of increased appetite and weight gain in cancer subjects with depression and nausea, as well as in non-depressed cancer patients, but there are not, as yet, randomized controlled trials showing its effect on cancer-associated anorexia-cachexia. The objective of this study is to evaluate the effect of mirtazapine as a pharmacological measure in the management of cancer-related anorexia-cachexia in patients in palliative care. A randomized, double-blind clinical trial involving 52 cancer patients with anorexia-cachexia in palliative care will be conducted. Patients will be randomized to receive mirtazapine or megestrol and will be evaluated longitudinally for a period of 8 weeks. After the initial evaluation and randomization, patients will be reassessed after 4 and 8 weeks at an outpatient clinic where they will be evaluated for the following variables: (1) General and demographic characteristics; (2) Usual food intake; (3) Anthropometric evaluation; (4) Presence and degree of symptoms using the Edmonton Symptom Assessment System; (4) Status performance using the Karnofsky performance status; (5) Quality of life using the QLQ-C30 Questionnaire; (6) Depression using the Hospital Anxiety and Depression Scale; (7) Prognosis using the Palliative Prognostic Score; (8) Evaluation of functional capacity using hand grip strength and gait speed; (9) Body composition using electrical bioimpedance and dual energy x-ray absorptiometry; (10) Physical Activity Behaviour using a tri-axial accelerometer. Patients will also be contacted via telephone calls at weeks 1, 2, 3, 5 and 6 for information regarding adverse events and drug compliance. The questioning about the occurrence of adverse events will also be performed at the outpatient clinic. Self-report of ingestion of tablets and counting of tablets on return of packages at the end of the study will be used to determine patient compliance. It is expect that use of mirtazapine can bring benefits increasing appetite and the body weight in cancer patientes in palliative care compared to the use of megestrol.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 50 years.
* Patients with confirmed diagnosis of cancer by histopathological examination, including those not yet submitted to any therapy because they are in the therapeutic definition phase and those whose therapies have already been suspended because they are ineffective.
* Patients with cancer progression, with either local or distant metastases, documented by radiological or histopathological methods.
* Patients complaining of anorexia graded by the patient as ≥ 5 by the Edmonton Sympton Assessement Scale.
* Patients with weight loss ≥ 2% in the last 2 months or weight loss ≥ 5% in the last 6 months, referred by the patient or documented in electronic medical records, compared to the stable weight before diagnosis.
* Patients with a life expectancy of ≥ 2 months by the Palliative Prognostic Score.
* Patients with performance status greater than or equal to 60% using the Karnofsky Performance Status scale.

Exclusion Criteria:

* Patients diagnosed with depression or using antidepressant therapy with a score ≥ 12 in the depression items of the Hospital Anxiety and Depression Scale.
* Patients with unstable doses of corticosteroids.
* Patients with moderate renal and/or hepatic dysfunction (total bilirubin ≥ 1.5x the upper limit of normal, AST and ALT ≥ 5x upper limit of normal or creatinine ≥1.5x upper limit of normal).
* Patients with Central Nervous System metastases.
* Patients with inability to take oral medications.
* Patients with mechanical obstruction of the gastrointestinal tract.
* Patients with clinically bulky ascites and generalized edema.
* Patients with reports of allergy to the medications studied.
* Patients with hypothyroidism with TSH levels greater than or equal to 5 μU/mL and free T4 less than 0.7 ng/dL.
* Patients with uncorrected hydroelectrolytic disturbances, with altered serum sodium, potassium and/ or ionic calcium.
* Patients with persistent and uncontrolled nausea and/or vomiting associated with gastrointestinal tract neoplasia and/or chemotherapeutic or radiotherapeutic treatment.
* Patients with pacemakers.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2022-02-02 (Actual); Study Completion 2022-02-02 (Actual)

PRIMARY OUTCOMES:
Change in appetite | 8 weeks
  Assessed by Edmonton Symptom Assessment Scale. This evaluation will be collected at baseline and after 8 weeks of follow-up. Changes in appetite will be divided into 3 categories according to the following definitions: appetite improvement will be a decrease ≥ 2 points in Edmonton Symptom Assessment Scale, maintenance of appetite as an improvement or worsening of 1 point and worsening of appetite as deterioration ≥ 2 points.
Change in body weight | 8 weeks
  Assessed by body weight. This evaluation will be collected at baseline and after 8 weeks of follow-up. The weight changes will be divided into 3 categories according to the following definitions: weight improvement will be a gain ≥ 1 kg, weight maintenance will be a loss < 500g or a gain < 1kg and weight loss will be a loss ≥ 500g.

SECONDARY OUTCOMES:
Change in body lean and fat mass | 8 weeks
  Assessed by body bioelectrical impedance and dual energy x-ray absorptiometry. They will be performed at baseline and after 8 weeks of follow-up. The body bioelectrical impedance will be performed using the ImpediMed DF50 mono-frequency system (ImpediMed Limited, Australia). The dual energy x-ray absorptiometry will be performed on the measuring table using the equipment-specific software.
Change in Quality of life | 8 weeks
  The European Organization for Research and Treatment of Cancer (EORTC) instrument QLQ-C30 Questionnaire will be used to assess quality of life at baseline and after 8 weeks of follow-up.
Assessment of muscle strength | 8 weeks
  Assessed by hand grip strenght measured by the use of a manual hydraulic dynamometer (Saehan, model SH 5.001, Koreia). It will be performed at baseline and after 8 weeks of follow-up.
Assessment of gait speed | 8 weeks
  The gait speed will be measured at 4 meters on usual speed. It will be performed at baseline and after 8 weeks of follow-up. The results will be expressed in m/s.
Physical Activity behaviour | 8 weeks
  Assessed by a tri-axial accelerometer to measure profile of spontaneous physical activity. It will be performed at first week and the last week of follow-up.
Incidence of treatment-related Adverse Events | 8 weeks
  Assessed by contact via telephone calls at weeks 1, 2, 3, 5 and 6 for information regarding treatment-related adverse events. The questioning about the occurrence of treatment-related adverse events will also be performed at the outpatient clinic at baseline and weeks 4 and 8 during the follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Nereida KC Lima, MD, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Clinics Hospital, Ribeirão Preto Medical School, University of São Paulo, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
IPD to be made available after the end of the study protocol.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: after the publication of the results of study.
Access Criteria: researchers after the review and approval of protocol by the principal investigator

REFERENCES:
- [Background] Riechelmann RP, Burman D, Tannock IF, Rodin G, Zimmermann C. Phase II trial of mirtazapine for cancer-related cachexia and anorexia. Am J Hosp Palliat Care. 2010 Mar;27(2):106-10. doi: 10.1177/1049909109345685. Epub 2009 Sep 23. PMID 19776373
- [Background] Theobald DE, Kirsh KL, Holtsclaw E, Donaghy K, Passik SD. An open-label, crossover trial of mirtazapine (15 and 30 mg) in cancer patients with pain and other distressing symptoms. J Pain Symptom Manage. 2002 May;23(5):442-7. doi: 10.1016/s0885-3924(02)00381-0. PMID 12007762
- [Background] Tomiska M, Tomiskova M, Salajka F, Adam Z, Vorlicek J. Palliative treatment of cancer anorexia with oral suspension of megestrol acetate. Neoplasma. 2003;50(3):227-33. PMID 12937858
- [Background] Wen HS, Li X, Cao YZ, Zhang CC, Yang F, Shi YM, Peng LM. Clinical studies on the treatment of cancer cachexia with megestrol acetate plus thalidomide. Chemotherapy. 2012;58(6):461-7. doi: 10.1159/000346446. Epub 2013 Feb 7. PMID 23406994
- See also: webpage of the Ribeirão Preto Medical School — http://fmrp.usp.br